CLINICAL TRIAL: NCT06448234
Title: Evaluating the Efficacy of AI-Guided vs. Standard Physician-Guided Dietary Supplement Prescriptions for Lowering LDL Cholesterol in Hypercholesterolemic Patients: A Randomized Controlled Pilot Trial
Brief Title: Evaluating the Efficacy of AI-Guided (GenAIS TM) vs. Standard Physician-Guided Dietary Supplement Prescriptions for Lowering LDL Cholesterol in Hypercholesterolemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW012
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hypercholesterolemia
Keywords: LDL cholesterol reduction; AI-guided prescriptions; Dietary supplements; Personalized nutrition
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants receive DS prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Interventions: Other: Standart supplementation therapy group
- AI-Guided Group (Experimental): Participants receive DS prescriptions determined by an AI system, which considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Interventions: Other: AI-guided supplementation therapy group

INTERVENTIONS:
Other: Standart supplementation therapy group — Participants receive supplement prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles
  Arms: Control Group
Other: AI-guided supplementation therapy group — Participants receive DS prescriptions determined by an AI system, which considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: AI-Guided Group

SUMMARY:
The trial compared AI-guided and standard physician-guided dietary supplement (DS) prescriptions for lowering LDL cholesterol (LDL-C) in hypercholesterolemic patients. The AI system used genetic, metabolic, and clinical data to personalize DS regimens, hypothesizing superior efficacy over traditional methods. This 3-month randomized, controlled trial involved adults aged 40-75 with specific LDL-C levels, excluding those with significant health risks. Participants were divided into a control group with physician-guided DS and an AI-guided group. The AI system from Triangel Scientific provided dynamic, personalized recommendations. Baseline and follow-up measurements included lipid profiles and adherence assessments. The AI-guided group showed significantly greater LDL-C reduction and improvement in other lipid markers. The study concluded that AI-guided DS prescriptions are more effective, suggesting a promising future for AI in personalized cholesterol management.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years.
* LDL-C level between 70 and 190 mg/dL, confirmed in at least two sequential checks conducted within the last six months prior to signing the consent form.

Exclusion Criteria:

* Personal history of cardiovascular disease or high risk (≥ 20%).

  * Triglycerides (TG) ≥ 400 mg/dL.
  * Body Mass Index (BMI) ≥ 35 kg/m²
  * Use of lipid-lowering drugs or supplements affecting lipid metabolism within the last three months.
  * Diabetes mellitus.
  * Known severe or uncontrolled thyroid, liver, renal, or muscle diseases.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
change in LDL-C | 180 days

SECONDARY OUTCOMES:
Percent change in high-sensitivity C-reactive protein ( | 180 days
Percent change in high-density lipoprotein cholesterol | 180 days
Percent change in total cholesterol. | 180 days
Percent change in serum triglycerides between the groups. | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

IPD SHARING:
Plan to Share IPD: Undecided